CLINICAL TRIAL: NCT01625572
Title: Ultrasound-assisted Bilateral Transversus Abdominis Plane Block for Open Prostatectomy
Acronym: TAPPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jurgen Birnbaum, PD Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAPPro
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Prostatectomy; Transversus Abdominis Plane Blockade; Pain
Keywords: general anaesthesia; epidural catheter; intravenous pain therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- general anesthesia and epidural catheter (control) (No Intervention): General anaesthesia
  * total intravenous anaesthesia with propofol 5-10 mg / kg / h,
  * remifentanil 0.1 to 0.3 micrograms / kg / min and muscle relaxation with cis-atracurium
  * use of a bispectral index
  * monitoring with a target range of 40-60
  * at the end of the anaesthesia all patients get 0.1 mg / kg morphine intravenously epidural catheter
  * plant of the epidural catheter under sterile conditions at the intervertebral space of the vertebral body 8-10 of the thoracic spine• local anaesthesia with lidocaine 1%
  * puncture with a Tuohy 18 G- needle, Lost of resistance technique
  * after a negative test dose with bupivacaine 0,5% isobar we inject fractional ropivacaine 10 ml 0,2%, after that continuous administration of ropivacaine 0,2% via patient-controlled-analgesia-device with a sweep rate of 6 ml/h, all Patients also receive an intravenous morphine-patient-controlled-analgesia-device
- general anesthesia and regional anesthesia (Experimental): General anesthesia
  * anesthesia with propofol 5-10 mg / kg / h, remifentanil 0.1 to 0.3 micrograms / kg / min and muscle relaxation with cis-atracurium
  * Bispektralindex monitoring with a target range of 40-60
  * at the end of the anesthesia all patients get 0.1 mg / kg morphine intravenously Transversus abdominis plane blockade
  * ultrasound visible needles, a special pin detection software
  * under visual control the needle moves into the space between Musculus obliquus internus and M. transversus abdominis
  * Under sonographic control we inject a local anesthetic depot (30 ml of ropivacaine 0.375%)
  * puncture is performed under constant protective nerve stimulation with a current of 1 mA, pulse duration 0.1 ms, frequency 2 Hz All Patients receive an i.v. Morphine-patient-controlled-analgesia-device
  Interventions: Procedure: Transversus abdominis plane blockade
- general anaesthesia and intravenous pain therapy (Experimental): General anaesthesia
  * total intravenous anesthesia with propofol 5-10 mg / kg / h, remifentanil 0.1 to 0.3 micrograms / kg / min and muscle relaxation with cis-atracurium
  * we use a of BIS monitoring with a target range of 40-60
  * at the end of the aneasthesia all patients get 0.1 mg / kg morphine intravenously intravenous pain therapy with
  * Morphine-patient-controlled-analgesia-device
  Interventions: Procedure: Morphine-patient-controlled-analgesia-device

INTERVENTIONS:
Procedure: Transversus abdominis plane blockade — Bilateral one time injection of local anaesthetic in the space between the transversus abdominis muscle and obliquus internus muscle preoperatively. Follow up for three days.
  Arms: general anesthesia and regional anesthesia
Procedure: Morphine-patient-controlled-analgesia-device — Morphine-patient-controlled-analgesia-device for three days: 1mg/ml, Dosage 2mg bolus injection on demand every 10 minutes possible.
  Arms: general anaesthesia and intravenous pain therapy

SUMMARY:
The purpose of this study is to compare the quality of a transversus abdominis plane blockade with an intravenous pain therapy with opioids. Due to the relatively low side effect profile and comparably few contraindications, this method offers a good option, to be a standard procedure or better alternative in the treatment of pain in surgery of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* patients at the age of 18 and above, who need an open prostatectomy
* written consent exists

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) classification > III
* Allergy to local anaesthesia
* Contraindications to one of the applied methods
* previous surgery on the abdominal wall
* chronic pain patients
* Myasthenia gravis
* alcohol dependence
* increased intraocular pressure
* lacking willingness to save and hand out data within the study
* Participation in another trial according to the German Drug Law
* accommodation in an institute due to an official or judicial order

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain in rest in the op-area | 3 days
  Pain in rest in the op-area during the first 3 days

SECONDARY OUTCOMES:
Opioid consumption | 3 days
  opioidconsumption during the first 3 days
Pain in motion in the op-area | 3 days
  Pain in the op-area in motion during the first three days
Pain outside the op-area | 3 days
  Pain outside the op-area during the first three days
Contentment with the pain therapy at all | 3 days
  Contentment with the pain therapy at all for the first three days
Frequency of postoperative vomiting and nausea | 3 days
  Frequency of postoperative vomiting and nausea during the first three days
Incidence of pruritus | 3 days
  Incidence of pruritus during the first three days
Tenesmuses of the bladder | 3 days
  Tenesmus of the bladder during the first three days
Contentment of the Patient at all | 3 days
  Contentment of the patient at all during the first three days

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Birnbaum, MD, Principal Investigator — Charite, Department of Anesthesiology and Intensive Care, Campus Mitte, Universitätsmedizin Berlin
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine Campus Charitè Mitte, Charite Universitätsmedizin Berlin, Berlin, State of Berlin, Germany